CLINICAL TRIAL: NCT04614636
Title: A Phase I, Open-Label, Multicenter Study of FT538 as Monotherapy in Relapsed/Refractory Acute Myelogenous Leukemia and in Combination With Monoclonal Antibodies in Relapsed/Refractory Multiple Myeloma
Brief Title: FT538 in Subjects With Advanced Hematologic Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated by the Sponsor.
Sponsor: Fate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FT538-101
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Acute Myeloid Leukemia; AML, Adult; Multiple Myeloma; Myeloma
Keywords: Acute Myeloid Leukemia; AML; Multiple Myeloma; daratumumab; elotuzumab; NK cell; cellular therapy; allogeneic cell therapy; allogeneic cellular therapy; CD38; Anti-CD38
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Cyclophosphamide; fludarabine; daratumumab; elotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- FT538 Monotherapy (Experimental): FT538 monotherapy in subjects with r/r AML
  Interventions: Drug: FT538; Drug: Cyclophosphamide; Drug: Fludarabine
- FT538 in Combination with Daratumumab (Experimental): FT538 in combination with daratumumab in subjects with r/r MM
  Interventions: Drug: FT538; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Daratumumab
- FT538 in Combination with Elotuzumab (Experimental): FT538 in combination with elotuzumab in subjects with r/r MM
  Interventions: Drug: FT538; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Elotuzumab

INTERVENTIONS:
Drug: FT538 — Experimental Interventional Therapy, Allogeneic Cell Therapy NK Cell
Drug: Cyclophosphamide — Lympho-conditioning Agent
Drug: Fludarabine — Lympho-conditioning Agent
Drug: Daratumumab — Monoclonal Antibody, CD38, Anti-CD38
  Other Names: Darzalex
  Arms: FT538 in Combination with Daratumumab
Drug: Elotuzumab — Monoclonal Antibody
  Other Names: Empliciti
  Arms: FT538 in Combination with Elotuzumab

SUMMARY:
This is a Phase I dose-finding study of FT538 as monotherapy in acute myeloid leukemia (AML) and in combination with monoclonal antibodies in multiple myeloma (MM). The study will consist of a dose-escalation stage and an expansion stage where participants will be enrolled into indication-specific cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of one of the following by treatment regimen:

   * Regimen A (FT538 monotherapy in r/r AML)

     * Primary refractory AML, or
     * Relapsed AML, defined as not in CR after one or more re-induction attempts; if >60 years of age, prior re-induction therapy is not required
   * Regimens B or C (FT538 + mAb in r/r MM)

     * Regimen B only: MM that has relapsed or progressed after at least two lines of therapies, including a proteasome inhibitor and an immunomodulatory drug
     * Regimen C only: MM that has relapsed or progressed after proteasome inhibitor therapy, and immunomodulatory therapy
     * Regimen B and Regimen C: Measurable disease as defined in the protocol
2. Capable of giving signed informed consent
3. Agreement to comply with study procedures as described in the Schedule of Activities
4. Agrees to contraceptive use as described in the protocol

Exclusion Criteria:

1. Females who are pregnant or breastfeeding
2. ECOG Performance Status ≥ 2
3. Evidence of insufficient hematologic function as defined in the protocol
4. Evidence of insufficient organ function defined as defined by the protocol
5. Clinically significant cardiovascular disease as defined by the protocol
6. Known active central nervous system (CNS) involvement by malignancy
7. Non-malignant CNS disease such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease or receipt of medications for these conditions in the 2-year period leading up to study enrollment
8. Currently receiving or likely to require systemic immunosuppressive therapy for any reason during the treatment period
9. Clinically significant infections including HIV, HBV and HCV
10. Live vaccine <6 weeks prior to start of lympho-conditioning
11. Receipt of an allograft organ transplant
12. Prior allogeneic HSCT or allogeneic CAR-T within 6 months of Day 1, or ongoing requirement for systemic graft-versus-host therapy
13. Known allergy to albumin (human) or DMSO
14. Presence of any medical or social issues that are likely to interfere with study conduct or may cause increased risk to subject
15. Any medical condition or clinical laboratory abnormality that per investigator or Medical Monitor judgement precludes safe participation in and completion of the study, or which could affect compliance with protocol conduct or interpretation of results

    Exclusion Criteria Specific to Regimen A (r/r AML)
16. Diagnosis of promyelocytic leukemia with t(15;17) translocation
17. Receipt of any biological therapy, chemotherapy, or radiation therapy, except for palliative purposes, within 2 weeks prior to Day 1 or five half-lives, whichever is shorter; or any investigational therapy within 28 days prior to Day 1

    Exclusion Criteria Specific to Regimens B and C (r/r MM)
18. Plasma cell leukemia defined as a plasma cell count >2000/mm3
19. Leptomeningeal involvement of MM
20. Receipt of any biological therapy, chemotherapy, or radiation therapy, except for palliative purposes, within 2 weeks prior to Day 1 or five half-lives, whichever is shorter; or any investigational therapy within 28 days prior to the first dose of mAb
21. Allergy or hypersensitivity to antibodies or antibody-related proteins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-10-17 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) within each dose level cohort | Cycle 1, Up to Day 29
Nature of dose-limiting toxicities within each dose level cohort | Cycle 1, Up to Day 29

SECONDARY OUTCOMES:
Incidence, nature, and severity of adverse events (AEs) of FT538 as monotherapy in r/r AML and in combination with daratumumab or elotuzumab in r/r multiple myeloma | Up to 5 years
Objective response rate (ORR) of FT538 as monotherapy in r/r AML and in combination with daratumumab or elotuzumab in r/r MM | From baseline tumor assessment up to approximately 2 years after last dose of FT538
  Proportion of subjects who achieve a CR, CRMRD-, CRi, MLFS, or PR, as determined by the investigator according to 2017 ELN criteria for AML, and the proportion of subjects with a best overall response of sCR, CR, VGPR, or PR, as determined by the investigator according to standard IMWG for MM response criteria
Duration of response (DOR) of FT538 in combination with daratumumab or elotuzumab in r/r MM | Up to 15 years
  Defined as the duration from the first occurrence of a documented objective response until the time of disease progression or relapse, or death due to progressive disease, as determined by the investigator according to standard IMWG response criteria
Progression-free survival (PFS) of FT538 in combination with daratumumab or elotuzumab in r/r MM | Up to 15 years
  Defined as the time from first dose of study treatment to disease progression or relapse, or to the day of death from any cause, as determined by the investigator according to standard IMWG response criteria
Relapse-free survival (RFS) of FT538 as monotherapy in r/r AML and in combination with daratumumab or elotuzumab in r/r MM | Up to 15 years
  Defined as the time from initial CR (including CRMRD-, CR, and CRi) to hematologic relapse or death due to any cause, as determined by the investigator according to 2017 ELN criteria for AML, and defined as the duration from the start of sCR or CR until the time of relapse from sCR or CR, as determined by the investigator according to standard IMWG response criteria for MM
Event-free survival (EFS) of FT538 as monotherapy in r/r AML | Up to 15 years
  defined as the time from first dose of lympho-conditioning to the date of PD, or relapse from CR or CRi, or death from any cause, according to 2017 ELN criteria
Overall survival (OS) of FT538 as monotherapy in r/r AML and in combination with daratumumab or elotuzumab in r/r MM | Up to 15 years
  defined as the time from first dose of lympho-conditioning to death from any cause
Time-to-best response of FT538 as monotherapy in r/r AML | Up to 15 years
  defined as the time from first dose of lympho-conditioning to best response
Determination of the pharmacokinetics (PK) of FT538 cells in peripheral blood | Study Days: 1, 2, 4, 8, 11, 15, 18, 22, 29
  The PK of FT538 in peripheral blood will be reported as the relative percentage of product (FT538) DNA versus patient DNA (% chimerism) measured from blood samples at the specified time points

CONTACTS AND LOCATIONS:
Overall Officials: Fate Trial Disclosure, Study Director — Fate Therapeutics, Inc
Locations (8):
- United States (8):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute at Tennessee Oncology, Nashville, Tennessee
  - St. David's South Austin Medical Center, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No